CLINICAL TRIAL: NCT00783848
Title: Validating PROMIS Instruments in Congestive Heart Failure Patients Receiving a Heart Transplant
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00009919; 5U01AR052186-02 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

The purpose of this research study is to learn about the experience and impact of having congestive heart failure (CHF). In particular, we hope to develop better questionnaires that can measure heart failure patients' quality-of-life.

DETAILED DESCRIPTION:
This project will assess the validity (including responsiveness) of selected Patient Reported Outcome Measurement Information System (PROMIS) instruments in patients with severe CHF who receive heart transplants. The following is a list of goals for this project:

* To estimate the responsiveness of PROMIS domain scores by comparing scores in patients with severe heart failure before and after a clinically significant event (heart transplant). The specific PROMIS domains assessed are physical functioning, fatigue, satisfaction with discretionary social activities, depression, and global health.
* To estimate the responsiveness of a disease-specific patient-reported outcome (PRO) measure, the Kansas City Cardiomyopathy Questionnaire (KCCQ), the Medical Outcomes Study Short Form-36 Vitality subscale (SF-36v2), and the Patient Health Questionnaire (PHQ-2).
* To collect cross-sectional and longitudinal data on traditional clinical measures of heart failure outcome (6-minute walk test and New York Heart Association [NYHA] class) that can inform the definition of a minimally important difference (MID) for the PROMIS domains of physical functioning, fatigue, satisfaction with discretionary social activities, depression, and global health.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure had to represent the greatest medical limitation on daily function for the patient in the judgment of the attending cardiologist
* Ability to read, write, and speak in English
* Ability to understand and provide informed consent
* Placement on heart transplant registry (awaiting heart transplant surgery)

Exclusion Criteria:

* Current diagnosis of psychosis or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through heart transplant program registries and in consultation with practicing cardiologists at Duke University, Stanford University, and the University of Pittsburgh.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the validity (including responsiveness) of selected PROMIS domains for patients with severe heart failure who receive a heart transplant. | baseline and 8-12 weeks post-transplant
  Clinical and patient-reported assessments will be performed at baseline and 8-12 weeks 86 (end of study). Clinical indicators of functioning will include the New York Heart 87 Association (NYHA) classification and the six-minute walk test. We will include the 88 Kansas City Cardiomyopathy Questionnaire (KCCQ), a disease-specific measure of health-89 related quality of life (HRQOL), as a point of reference for understanding the relative 90 validity (including responsiveness) of the PRPROMIS item banks. Instruments will include 91 PROMIS computerized adaptive tests (CATS).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Weinfurt, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania